CLINICAL TRIAL: NCT01581515
Title: 2-phased Randomized Comparison Between PromusTMElementTM Versus Xience PRIME® Stent
Brief Title: Assessment of Stent Malapposition and Neointimal Coverage on Optical coHerence Tomography at Post-procedure and 3 Months After Platinum Chromium Alloy Of the Element™ Stent Implantation
Acronym: ANCHOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Myeong-Ki Hong, MD, Ph D, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2011-0080
Record Dates: First submitted 2012-04-11; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P-E group (Active Comparator): Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; either Promus Element or Xience Prime
  Interventions: Device: Promus Element everolimus eluting coronary stent
- X-P group (Active Comparator): Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; either Promus Element or Xience Prime
  Interventions: Device: Xience Prime everolimus eluting coronary stent

INTERVENTIONS:
Device: Promus Element everolimus eluting coronary stent — Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; either Promus Element or Xience Prime
  Arms: P-E group
Device: Xience Prime everolimus eluting coronary stent — Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; either Promus Element or Xience Prime
  Arms: X-P group

SUMMARY:
The purpose of this study is to compare the degree of stent malapposition on an immediate optical coherence tomography (OCT) after nominal stent pressure and at a final post-procedure OCT (ANCHOR-I) and the neointimal coverage on 3-months OCT following the intervention with the randomly assigned two drug-eluting stents (DES), PromusTMElementTM stents versus Xience PRIME® stents.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 20 years old
* Significant coronary de novo lesion (> 70% by quantitative angiographic analysis) treated by single DES in each vessel.
* Patients with stable angina who are considered for coronary revascularization with stent implantation.
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Complex lesion morphologies such as aorto-ostial, unprotected left main, chronic total occlusion, graft, thrombosis, and restenosis
* Reference vessel diameter < 2.5 mm or > 4.0mm and lesion length > 28 mm
* Heavy calcified lesions (definite calcified lesions on angiogram)
* Lesions requiring more than 2 DES in each vessel
* Acute coronary syndrome
* Contraindication to anti-platelet agents
* Treated with any DES within 3 months at other vessel
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy 1 year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
the ratio of the malapposed strut | Participants will be followed from first OCT invervention to 3month OCT following intervention
  The ratio of the malapposed strut, on an immediate OCT after nominal stent pressure and at a final post-procedure between two different DES; ANCHOR-I

SECONDARY OUTCOMES:
Incidence of stent malapposition | 3months OCT following intervention
Neointimal coverage(ANCHOR II) | 3 month-OCT after stent implantation
Incidence of plaque prolapse | final postprocedural OCT
Evaluation of stent expansion | an immediate and post-procedural OCT
Stent malapposition | on 3 month OCT intervention

CONTACTS AND LOCATIONS:
Overall Officials: Myeong-Ki Hong, MD.PhD., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu/Sinchon-dong, South Korea

REFERENCES:
- [Derived] Kim BK, Shin DH, Kim JS, Ko YG, Choi D, Jang Y, Hong MK. Randomized comparison of acute stent malapposition between platinum-chromium versus cobalt-chromium everolimus-eluting stents. Int J Cardiovasc Imaging. 2015 Feb;31(2):269-77. doi: 10.1007/s10554-014-0557-y. Epub 2014 Oct 28. PMID 25345751